CLINICAL TRIAL: NCT04721964
Title: Evaluation of the Effects of Routine Iron Supplementation in Children on Gastrointestinal Iron Losses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Principal Investigator, Nicole Stoffel, Principal Investigator, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FeLo
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Iron Deficiency Anemia; Gastro Intestinal Bleeding; Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Gastrointestinal Hemorrhage | interventions — ferric ammonium citrate

STUDY DESIGN:
Intervention Model Description: Prospective intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All 24 participants will daily consume 6 mg iron/kg body weight for 13 weeks to correct their anaemia and increase their iron stores.
  Interventions: Dietary Supplement: Ferric ammonium citrate and ferrous fumarate syrup (Ranbaxy Ranferon-12 Syrup, Ranbaxy Laboratories, Gurgaon, India)

INTERVENTIONS:
Dietary Supplement: Ferric ammonium citrate and ferrous fumarate syrup (Ranbaxy Ranferon-12 Syrup, Ranbaxy Laboratories, Gurgaon, India) — Daily supplementation with iron syrup for 13 weeks. The dosage will be calculated based on body weight and adjusted after 4 and 8 weeks of intervention

SUMMARY:
Iron deficiency anaemia (IDA) is common among infants and young children in sub-Saharan Africa.Oral iron administration is usually recom-mended as cost effective measure to prevent and treat iron deficiency (ID) and IDA during childhood. In Kenya, national nutrition policies for anaemia prevention recommend a daily dose of 3-6 mg ele-mental iron per kg body weight if a child is diagnosed with anaemia.

Using a novel technology, recent research found increased iron losses during iron supplementation. In an explorative analysis of stool samples collected from Gambian toddlers (Speich et al., 2020), an increase in faecal iron losses during iron supplementation was reported. The present study is aiming to analyse a relationship between routine iron supplementation and increased faecal occult blood losses in 24 Kenyan children with anaemia and iron deficiency in a more structured manner.

Secondary objectives of the study are to measure and monitor iron and inflammatory status during the course of the study and to quantify long-term iron absorption and iron losses during a 12-weeks iron supplementation period, in order to put iron balance into relationship to occurring faecal occult blood losses during such an intervention.

DETAILED DESCRIPTION:
Infants and young children in sub-Saharan Africa have high rates of iron deficiency anaemia (IDA), which adversely affects their growth and cognitive development. WHO recommends daily administration of 3 mg elemental iron per kg body weight in form of drops or syrup in 6-23 month-old ID or anaemic infants. In settings where anaemia prevalence in this age group is >40%, WHO further recommends daily administration of 10-12.5 mg elemental iron for prevention of ID and anaemia. The Kenyan Ministry of Health adopted the WHO strategy to treat IDA in its "Basic Paediatric Protocols" released in 2016, and specified a dose of 3-6 mg elemental Fe per kg body weight and day.

WHO guidelines for anaemia prevention and control in infants aged 6-23 months are based on a systematic review and meta-analysis of randomized controlled trials investigating the effect of daily iron supplementation on health in infants. The review reported a significantly lower risk of iron-deficiency anaemia in infants when supplemented. However, iron supplements and iron-containing micronutrient powders (MNPs) do not always show efficacy; for example, in a recent large intervention trial in Pakistan, there was no significant effect of 12 months of iron supplementation on haemoglobin status.

Among the many potential factors contributing to the limited success of health and nutrition policies in reducing the prevalence of iron deficiency, increased iron losses during iron supplementation have not been considered. In a recent study in Gambian toddlers, a 3.4-fold increase in iron losses was detected, specifically from 0.22 (0.19;0.29) mg/d to 0.75 (0.55;0.87) mg/d, during a 12-week iron intervention with daily consumption of 12 mg iron as ferrous fumarate in MNPs routinely distributed by the United Nations Children's Fund and the World Food Program. Furthermore, the administered iron dose significantly correlated with faecal haemoglobin concentration in the Gambian toddlers. In a recent iron supplementation pilot study in Kenyan toddlers, the investigators measured a significant increase in faecal haemoglobin concentration during iron supplementation. Increased basal iron losses during iron supplementation could also be detected in 10 Swiss women. Several endoscopy studies have suggested iron supplementation may cause irritation/inflammation of the gut mucosa, potentially leading to gastrointestinal blood losses.

To explore a potential relationship between iron supplementation with common iron supplements and increased faecal occult (small traces of blood, not visible in stool) blood losses, this study will measure haemoglobin and porphyrin content in stool samples collected before and throughout a 91-day iron supplementation intervention. Intervention product will be 6 mg iron / kg body weight as ferric ammonium citrate and ferrous fumarate syrup (Ranbaxy Ranferon-12 Syrup, Ranbaxy Laboratories, Gurgaon, India) administered daily. Faecal occult blood losses will also be compared to absolute iron losses determined by the recently developed dilution of stable iron isotopes methodology. The study population will consist of 24 anaemic 2-years old children in Kwale County of southern coastal Kenya. The hypothesis of the investigators is that iron status will improve, but faecal occult blood losses will increase. The data from this project may provide valuable information towards the development of safer and more effective iron supplementation regimens.

ELIGIBILITY:
Inclusion Criteria:

* Participation in former Fe_HMO_GOS study (JKUAT/IERC No. 301019) or INSPIRE study (JKUAT/IERC No. JKU/2/4/896B).
* Mildly to moderately anaemic defined as 9.0 g/dL ≤ Hb < 11 g/dL.
* Iron deficiency defined as ZPP >80μmol/mol.
* Willingness of the caregiver to participate in the study.
* Residence in the study area for the period of the study.
* The informed consent form has been read and signed by the participant's caregiver (or has been read out to the participant's caregiver in case of illiteracy)
* Assessment of good health by professional staff at Msambweni District Hospital.

Exclusion Criteria:

* Hb <9 g/L or >11 g/L.
* Zinc ProtoPorphyrin ≤80 μmol/mol.
* Severe underweight (Z-score weight-for-age ≤-3).
* Severe wasting (Z-score weight-for-height ≤-3).
* Antibiotics consumption in the 7 days prior to screening.
* Consumption of iron supplements in the 14 days prior to screening.
* Any severe metabolic, gastrointestinal, kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the guardian's statement or medical examination (health booklet)).
* Participants taking part in other studies requiring the drawing of blood or involving medical or physical interventions.

Ages: 23 Months to 29 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Fecal occult blood concentration | Day 4-7 (baseline)
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Fecal occult blood concentration in the samples will be estimated from haemoglobin and porphyrin content in stool samples. These measurements will be assessed from stool aliquots, that will be shipped frozen to Mayo Clinic Laboratory (Rochester, USA), using highly specific hemoquant assay.
Fecal occult blood concentration | Day 32-35
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Fecal occult blood concentration in the samples will be estimated from haemoglobin and porphyrin content in stool samples. These measurements will be assessed from stool aliquots, that will be shipped frozen to Mayo Clinic Laboratory (Rochester, USA), using highly specific hemoquant assay.
Fecal occult blood concentration | Day 60-63
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Fecal occult blood concentration in the samples will be estimated from haemoglobin and porphyrin content in stool samples. These measurements will be assessed from stool aliquots, that will be shipped frozen to Mayo Clinic Laboratory (Rochester, USA), using highly specific hemoquant assay.
Fecal occult blood concentration | Day 95-98
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Fecal occult blood concentration in the samples will be estimated from haemoglobin and porphyrin content in stool samples. These measurements will be assessed from stool aliquots, that will be shipped frozen to Mayo Clinic Laboratory (Rochester, USA), using highly specific hemoquant assay.

SECONDARY OUTCOMES:
Iron status: Hemoglobin (g/dl) (Hb) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. Hb concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Zinc protoporphyrin (µmol/mol) (ZPP) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. ZPP concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Soluble Transferrin Receptor (mg/L) (sTfR) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of sTfR concentration.
Iron status: Serum Ferritin (ug/L) (SF) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of SF concentration.
Iron status: Serum Hepcidin (nM) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit.1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland, for analysis of serum hepcidin.
Iron status: Hemoglobin (g/dl) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. Hb concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Zinc protoporphyrin (µmol/mol) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. ZPP concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Soluble Transferrin Receptor (mg/L) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of sTfR concentration.
Iron status: Serum Ferritin (ug/L) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of SF concentration.
Iron status: Serum Hepcidin (nM) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit.1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland, for analysis of serum hepcidin.
Iron status: Hemoglobin (g/dl) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. Hb concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Zinc protoporphyrin (µmol/mol) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. ZPP concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Soluble Transferrin Receptor (mg/L) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of sTfR concentration.
Iron status: Serum Ferritin (ug/L) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of SF concentration.
Iron status: Serum Hepcidin (nM) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit.1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland, for analysis of serum hepcidin.
Iron status: Hemoglobin (g/dl) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. Hb concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Zinc protoporphyrin (µmol/mol) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. ZPP concentration will be measured immediately after blood withdrawal using an iCheck Anaemia diagnostic device (BioAnalyt GmbH, Teltow, Germany).
Iron status: Soluble Transferrin Receptor (mg/L) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of sTfR concentration.
Iron status: Serum Ferritin (ug/L) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quatification of SF concentration.
Iron status: Serum Hepcidin (nM) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit.1 mL full blood samples will then be aliquoted and the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland, for analysis of serum hepcidin.
Inflammation status: alpha Glycoprotein (g/L) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of AGP.
Inflammation status: C-reactive protein (mg/L) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of CRP.
Inflammation status: Fatty Acids Binding Protein (ng/ml) | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland.
  I-FABP concentrations will be analysed after completion of the study at the ETH laboratory, using commercially available ELISA kits.
Inflammation status: C-reactive protein (mg/L) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of CRP.
Inflammation status: alpha Glycoprotein (g/L) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of AGP.
Inflammation status: Fatty Acids Binding Protein (ng/ml) | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland.
  I-FABP concentrations will be analysed after completion of the study at the ETH laboratory, using commercially available ELISA kits.
Inflammation status: C-reactive protein (mg/L) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of CRP.
Inflammation status: alpha Glycoprotein (g/L) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of AGP.
Inflammation status: Fatty Acids Binding Protein (ng/ml) | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland.
  I-FABP concentrations will be analysed after completion of the study at the ETH laboratory, using commercially available ELISA kits.
Inflammation status: C-reactive protein (mg/L) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of CRP. .
Inflammation status: alpha Glycoprotein (g/L) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. A serum aliquot of only 100-200 μL will be analysed externally in the VitMin Lab, Willstaett, Germany, using a multiplex ELISA assay developed by Erhardt et al. (Erhardt et al., 2004) for quantification of AGP.
Inflammation status: Fatty Acids Binding Protein (ng/ml) | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. After aliquotting 1 mL full blood samples, the remaining blood samples will be centrifuged, all serum aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland.
  I-FABP concentrations will be analysed after completion of the study at the ETH laboratory, using commercially available ELISA kits.
Red Blood Cells isotopic composition | Baseline (day 7)
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will be aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. For iron isotopic composition each blood sample will be analysed in duplicate under chemical blank monitoring. Whole blood samples will be mineralised using an HNO3 and microwave digestion. This is followed by a separation of the sample matrix by anion-exchange chromatography and a subsequent precipitation step with ammonium hydroxide. The isotopic analyses will be performed by inductively coupled plasma mass spectrometry (ICPMS) using a high resolution double focusing mass spectrometer equipped with a multi-collector system for simultaneous ion beam detection.
Red Blood Cells isotopic composition | Day 35
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will be aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. For iron isotopic composition each blood sample will be analysed in duplicate under chemical blank monitoring. Whole blood samples will be mineralised using an HNO3 and microwave digestion. This is followed by a separation of the sample matrix by anion-exchange chromatography and a subsequent precipitation step with ammonium hydroxide. The isotopic analyses will be performed by inductively coupled plasma mass spectrometry (ICPMS) using a high resolution double focusing mass spectrometer equipped with a multi-collector system for simultaneous ion beam detection.
Red Blood Cells isotopic composition | Day 63
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will be aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. For iron isotopic composition each blood sample will be analysed in duplicate under chemical blank monitoring. Whole blood samples will be mineralised using an HNO3 and microwave digestion. This is followed by a separation of the sample matrix by anion-exchange chromatography and a subsequent precipitation step with ammonium hydroxide. The isotopic analyses will be performed by inductively coupled plasma mass spectrometry (ICPMS) using a high resolution double focusing mass spectrometer equipped with a multi-collector system for simultaneous ion beam detection.
Red Blood Cells isotopic composition | Day 98
  Venipuncture blood withdrawal (3 mL) will be performed at each hospital visit. 1 mL full blood samples will be aliquoted and stored at -20°C at the study site until all samples will be shipped frozen to ETH Zurich, Switzerland. For iron isotopic composition each blood sample will be analysed in duplicate under chemical blank monitoring. Whole blood samples will be mineralised using an HNO3 and microwave digestion. This is followed by a separation of the sample matrix by anion-exchange chromatography and a subsequent precipitation step with ammonium hydroxide. The isotopic analyses will be performed by inductively coupled plasma mass spectrometry (ICPMS) using a high resolution double focusing mass spectrometer equipped with a multi-collector system for simultaneous ion beam detection.
Fecal calprotectin concentration | Day 4-7 (baseline)
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Stool aliquots will be shipped frozen to ETH Zurich, Switzerland, for determination of calprotectin content using commercially available calprotectin kits.
Fecal calprotectin concentration | Day 32-35
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Stool aliquots will be shipped frozen to ETH Zurich, Switzerland, for determination of calprotectin content using commercially available calprotectin kits.
Fecal calprotectin concentration | Day 60-63
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Stool aliquots will be shipped frozen to ETH Zurich, Switzerland, for determination of calprotectin content using commercially available calprotectin kits.
Fecal calprotectin concentration | Day 95-98
  72 h stool samples will be collected from the study participants during 4 collection periods (day 4-7 (baseline), day 32-35, day 60-63, day 95-98). Stool aliquots will be shipped frozen to ETH Zurich, Switzerland, for determination of calprotectin content using commercially available calprotectin kits.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole U Stoffel, PhD, Principal Investigator — ETH
Locations (1):
- Msambweni County Referral Hospital, Mombasa, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Speich C, Wegmuller R, Brittenham GM, Zeder C, Cercamondi CI, Buhl D, Prentice AM, Zimmermann MB, Moretti D. Measurement of long-term iron absorption and loss during iron supplementation using a stable isotope of iron (57 Fe). Br J Haematol. 2021 Jan;192(1):179-189. doi: 10.1111/bjh.17039. Epub 2020 Aug 30. PMID 32862453
- [Derived] Giorgetti A, Nyilima S, Stoffel NU, Moretti D, Mwasi E, Karanja S, Zeder C, Speich C, Netland C, Jin Z, Zimmermann MB, Brittenham GM. Stable iron (58Fe) isotopic measurements in Kenyan toddlers during 3 months of iron supplementation demonstrate that half of the iron absorbed is lost. Br J Haematol. 2024 May;204(5):2057-2065. doi: 10.1111/bjh.19319. Epub 2024 Feb 1. PMID 38302093